CLINICAL TRIAL: NCT01678040
Title: MRI Assessment of the Effect of Preload on Ventricular Volumes and Function in Healthy Adult Volunteers
Brief Title: Ventricular Volume as Assessed by Cardiac Magnetic Resonance
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Lars Grosse-Wortmann, Staff Cardiologist, The Hospital for Sick Children
Other Study IDs: 1000031585
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Arrhythmogenic Right Ventricular Cardiomyophathy (ARVC)
Keywords: Ventricular Volume; Cardiac Magnetic Resonance; Echocardiogram

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac Magnetic Resonance: The CMR examinations will be performed in the cardiac MRI scanner (Siemens "Avanto", 1.5 Tesla, Erlangen, Germany) at the Hospital for Sick Children. A brief echocardiogram will be performed using a GE Vivid 7 or Vivid E9 machine (General Electric Medical Systems, Wisconsin, USA) We will image from standard parasternal long axis and apical four-chamber before and after completed hydration.

SUMMARY:
One of the many uses of cardiac magnetic resonance (CMR) is the assessment of right ventricular (RV) volumes. There are a number of congenital heart defects and acquired conditions in which management decisions are fundamentally based on ventricular volumes. The "gold standard" for assessment of RV volume is CMR. It has better near-field resolution than echo and excellent contrast between the blood pool and the myocardium. CMR is more suitable to the irregular geometry of the RV. The objectives of this study are (1) to assess ventricular volumes in the fasting state and after oral hydration in order to assess the effect of fluid status on ventricular volumes as measured by CMR; (2) to evaluate the effect of hydration on ventricular volumes compared the effect of with inter-observer and intra-observer variability, and; (3) to evaluate the effects of chamber volume on chamber deformation, including strain and peak strain rate. This study hypothesizes that (1) hydration status has an effect on right and left heart volumes, measured by CMR in healthy volunteers; (2) the effect of volume status will be a more significant contributor to variability in RV volumetry than that of inter-observer variability and intra-observer variability, and; (3) atrial and Ventricular deformation corrected for chamber size or volume is more accurate than when uncorrected for volume.

DETAILED DESCRIPTION:
1. To assess ventricular volumes in the fasting state and after oral hydration in order to assess the effect of fluid status on ventricular volumes as measured by CMR.
2. To evaluate the effect of hydration on ventricular volumes compared the effect of with inter-observer and intra-observer variability.
3. To evaluate the effects of chamber volume on chamber deformation, including strain and peak strain rate.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be healthy

Exclusion Criteria:

* Individuals who are unable to participate in an overnight fast will be excluded
* Those with known or suspected structural heart disease will be excluded
* A screening form to identify pre-existing cardiac conditions will be completed by the subject prior to participation in this study. If a pre-existing condition cardiac condition is identified, or suspected they will be excluded from the study.
* If any functional abnormality is detected at any stage by echocardiography or by CMR the study will be terminated. Common anatomical variants, which are generally regarded as normal variants (such as a patent foramen ovale, or a persistent left superior vena cava) will not lead to exclusion from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Staff from the Heart Centre at The Hospital for Sick Children will be sent an email notifying them of the study. They will be invited to obtain the particulars of the study by replying to Dr. Daryl Schantz or Dr. Lars Grosse-Wortmann. If they agree to participate Dr. Schantz will obtain written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Fluid Status | Day 1
  To assess ventricular volumes in the fasting state and after oral hydration in order to assess the effect of fluid status on ventricular volumes as measured by CMR.

SECONDARY OUTCOMES:
Hydration | Day 1
  To evaluate the effect of hydration on ventricular volumes compared the effect of with inter-observer and intra-observer variability.
Chamber Deformation | Day 1
  To evaluate the effects of chamber volume on chamber deformation, including strain and peak strain rate

CONTACTS AND LOCATIONS:
Overall Officials: Lars Grosse-Wortmann, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada